CLINICAL TRIAL: NCT04517175
Title: Could Ki-67 be Used as a Diagnostic or Prognostic Marker in Hemato-oncological Diagnostics?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University (Other)
Collaborators: Zuyderland Medisch Centrum (Other); Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Stefan Mestrum, Principal Investigator, Maastricht University
Other Study IDs: 2019-1345
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Myelodysplastic Syndrome/Neoplasm
Keywords: Ki-67
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Myelodysplastic syndrome (MDS) patients: MDS patients will be divided according to prognostic parameters in sub-cohorts.
  Interventions: Diagnostic Test: Flow cytometry
- Acute myeloid Leukemia (AML) patients: AML patients will be divided according to prognostic parameters in sub-cohorts.
  Interventions: Diagnostic Test: Flow cytometry
- Myelodysplastic syndrome/neoplasm (MDS/MPN) patients: MDS/MPN patients will be divided according to prognostic parameters in sub-cohorts.
  Interventions: Diagnostic Test: Flow cytometry

INTERVENTIONS:
Diagnostic Test: Flow cytometry — Flow cytometric immunophenotyping and determination of proliferative activity by means of Ki-67.

SUMMARY:
Ki-67 is used as a marker for determination of the proliferative activity in solid tumors. The use within hemato-oncological malignancies is limited. This is related to limited technical possibilities of flow cytometry in the past. Meanwhile, flow cytometry in hemato-oncological malignancies has progressed to assessment of 8 colors and makes it possible to add Ki-67 as an additional marker to the 8-color panels. Adding Ki-67 to these panels could lead to improved diagnosis and prediction of therapy response for a number of hemato-oncological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* MDS and AML patients

Exclusion Criteria:

* Ongoing radio- and/or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in which a hemato-oncological malignancy is found and are at least 18 years old. These patients can be male and female.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Maturation patterns diagnosis | 5 years
  Maturation patterns based on immunophenotype for red blood cells and several types of immune cells and their respective contributions to diagnosis.
  Maturation patterns are scored by various methods/combinations to form diagnostic score. A higher diagnostic score will lead to a more likely diagnose for MDS and/or AML.
Proliferative index diagnosis | 5 years
  Ki-67 proliferative index (within populations and maturation) and its contribution to diagnosis. A lower Ki-67 proliferative index will lead to a more likely diagnose for MDS and/or AML.
Proliferative index prognosis | 5 years
  Ki-67 as prognostic parameter. A lower Ki-67 proliferative index will (hypothetically) lead to worse prognosis for MDS and AML in terms of: transfusion dependence (expressed in amount of transfusions in 2 months), chemotherapy response (expressed as total remission, normalization of blood values, possibly also normalization of cytogenetics in bone marrow cells), overall survival (expressed in months after diagnosis), Risk scores. Higher risk scores are correlated with worse prognosis.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nies KPH, Kraaijvanger R, Lindelauf KHK, Drent RJMR, Rutten RMJ, Ramaekers FCS, Leers MPG. Determination of the proliferative fractions in differentiating hematopoietic cell lineages of normal bone marrow. Cytometry A. 2018 Nov;93(11):1097-1105. doi: 10.1002/cyto.a.23564. Epub 2018 Sep 3. PMID 30176186